CLINICAL TRIAL: NCT03502161
Title: Clinical Evaluation of the QuantiFERON CMV Assay
Status: Terminated | Type: Observational
Why Stopped: Business decision.
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C16-CMV-001
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: CMV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: Those receiving a SOT and coming off either 3 months or 6 months of antiviral prophylaxis.
  Interventions: Device: QuantiFERON CMV Assay

INTERVENTIONS:
Device: QuantiFERON CMV Assay — Assay to measure cell-mediated immune function using QuantiFERON CMV assay.

SUMMARY:
Validate the use of the device in the clinical setting for assessing the risk of CMV Infection in SOT recipients after the completion of antiviral prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Adult CMV D+/R- liver, kidney, heart, pancreas, lung, intestinal, or combined transplant recipients that are 18 years of age or older.
* Scheduled to receive between 3 to 6 months of antiviral prophylaxis
* Provide Informed Consent

Exclusion Criteria:

* Subjects less than 18 years old
* Scheduled to receive longer than 6 months or shorter than 3 months of prophylaxis
* Unable to provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CMV D+/R- SOT recipients older than 18 that are receiving 3-6 months of antiviral prophylaxis and can provide Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in time to CMV Infection between sub-groups of QF-CMV assay classifications. | At time of prophylaxis termination, +1 month from termination, +2 months from termination
  Measurement of QF-CMV result

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tolkoff-Rubin N, Rubin R. The impact of cytomegalovirus infection on graft function and patient outcome. Graft 1999; 2:S101-3.
- [Background] Singh N. Preemptive therapy versus universal prophylaxis with ganciclovir for cytomegalovirus in solid organ transplant recipients. Clin Infect Dis. 2001 Mar 1;32(5):742-51. doi: 10.1086/319225. Epub 2001 Feb 20. PMID 11229841